CLINICAL TRIAL: NCT05101837
Title: Feasibility and Effectiveness of a Specific App to Delivery Mindfulness Sessions to Patients with Different Kinds of Pain Condition: a Pilot Study
Brief Title: Feasibility and Effectiveness of a Specific App to Delivery Mindfulness Sessions
Acronym: BE_BI_MIND_APP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BE_BI_MIND_APP
Record Dates: First submitted 2021-09-27; First posted 2021-11-01 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Migraine; Neuropathic Pain
MeSH Terms: conditions — Migraine Disorders; Neuralgia

STUDY DESIGN:
Intervention Model Description: independent interventional non pharmacological pilot study with APP for mindfulness practice on android
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MIND-GROUP (Experimental): Daily mindfulness sessions on android
  Interventions: Device: Home program

INTERVENTIONS:
Device: Home program — Regular mindfulness guided face-to-face program, by using the technology with android to receive mindfulness sessions for daily practice and to assess the feasibility and the effectiveness of behavioural approach base on mindfulness delivered with this modality

SUMMARY:
A standardized behavioural approach based on mindfulness delivered mainly by a specific APP on android will be developed and applied for patients with chronic pain conditions, as migraine and neuropathic pain.

The aim of this pilot study:

The investigators propose a pilot study to enforce the application of a Home-program for patients with different pain conditions, to learn mindfulness practice, added to a regular mindfulness guided face-to-face program, by using the technology with android to receive mindfulness sessions for daily practice and to assess the feasibility and the effectiveness of behavioural approach base on mindfulness delivered with this modality.

DETAILED DESCRIPTION:
Background and significance Different clinical experiences confirmed the effectiveness of interventions based on the application of standardized behavioural approaches to support pharmacological traditional treatments for pain conditions in the last decades. Also, different clinical experiences were performed by using electronic devices to deliver home-sessions of behavioral approach (mindfulness) to patients that can practice regularly and supported by mindfulness recorded sessions

The aspect of feasibility of these treatments is not reported in published studies, but it can be estimated that standardized behavioural therapies are used in helping patients to obtain a better outcome for pain management

In particular, the use of technology to deliver behavioral exercises to patients suffering from different pain conditions, as neuropathic pain and migraine, have been reported in the literature of the last decades. Exercise-based on telemedicine and smartphone applications seem appropriate, as they have been recently tested in the management of chronic pain conditions to reinforce the efficacy of pharmacological therapies and to teach patients to manage their pain and to be more conscious about their clinical condition and about the use of drugs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Neuropathic Pain and Chronic Migraine
* written informed consent

Exclusion Criteria:

* co-existent severe medical or psychiatric illnesses, documented by specific previous diagnoses
* seizures
* use of opioids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Adherence at the program | 2 months
  To test the adherence of patients at the program. This evaluation will be conducted at the end of the program (Morisky, 2008)

SECONDARY OUTCOMES:
Monthly headache days or days with pain and medication intake | at 2 months
  Changes in monthly headache days or days with pain and medication intake compared with baseline, by daily diary card to record pain level on a Visual Analogue Scale (VAS) from 0 as no pain to 10 as Maximum pain; also medication intake reporded on the daily diary card.
Self-efficacy | at 2 months
  Changes in self-efficacy (by GSE score) (Generalized Self-Efficacy Scale) at 2months from the beginning of the program compared to baseline (minimum score 10-low level of self- efficacy=worse outcome; maximum score 40-high level of self-efficacy=better outcome ) (Scholz, 2002)
FIVE FACET MINDFULNESS | at 2 months
  Changes in FFMQ questionnaire FIVE FACET MINDFULNESS QUESTIONNAIRE compared to baseline (Baer, 2006): this questionnaire measures the mindfulness ability of patients before and after the APP application.
  (minimum score 113.7-low mindfulness ability=worse outcome ; maximum score 144.3-high mindfulness ability=better outcome)
System Usability Scale | up to 2 months
  Changes in SUS scale (System Usability Scale) at the end of the program (Brooke, 1996): this scale measures the usability of the APP.
  (minimum score 0-low usability of the APP=worse outcome; maximum score 100-high usability of the APP=better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adamse C, Dekker-Van Weering MG, van Etten-Jamaludin FS, Stuiver MM. The effectiveness of exercise-based telemedicine on pain, physical activity and quality of life in the treatment of chronic pain: A systematic review. J Telemed Telecare. 2018 Sep;24(8):511-526. doi: 10.1177/1357633X17716576. Epub 2017 Jul 11. PMID 28696152
- [Background] Alexander JC, Joshi GP. Smartphone applications for chronic pain management: a critical appraisal. J Pain Res. 2016 Sep 26;9:731-734. doi: 10.2147/JPR.S119966. eCollection 2016. No abstract available. PMID 27713649
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Friedman DI, Rajan B, Seidmann A. A randomized trial of telemedicine for migraine management. Cephalalgia. 2019 Oct;39(12):1577-1585. doi: 10.1177/0333102419868250. Epub 2019 Aug 26. PMID 31450969
- [Background] Rizzoli PB, Grazzi L. Adaptation of the management of chronic migraine patients with medication overuse to the suspension of treatment protocols during the COVID-19 pandemic: Lessons from a tertiary headache center in Milan-6-month results. Headache. 2021 Jun;61(6):961-962. doi: 10.1111/head.14140. Epub 2021 Jun 21. No abstract available. PMID 34153116
- [Background] Linardon J. Can Acceptance, Mindfulness, and Self-Compassion Be Learned by Smartphone Apps? A Systematic and Meta-Analytic Review of Randomized Controlled Trials. Behav Ther. 2020 Jul;51(4):646-658. doi: 10.1016/j.beth.2019.10.002. Epub 2019 Nov 26. PMID 32586436
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Qubty W, Patniyot I, Gelfand A. Telemedicine in a pediatric headache clinic: A prospective survey. Neurology. 2018 May 8;90(19):e1702-e1705. doi: 10.1212/WNL.0000000000005482. Epub 2018 Apr 6. PMID 29626180
- [Background] Rosser BA, Eccleston C. Smartphone applications for pain management. J Telemed Telecare. 2011;17(6):308-12. doi: 10.1258/jtt.2011.101102. Epub 2011 Aug 15. PMID 21844177